CLINICAL TRIAL: NCT06283875
Title: A Prospective, Single Center Clinical Study on the Clinical Significance of Personalized ctDNA-MRD in Predicting the Efficacy and Monitoring the Risk of Recurrence of Cervical Cancer
Brief Title: The Exploration of Personalized ctDNA Based MRD in the Clinical Significance of Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROMISEPLUS-301
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Cancer
Keywords: ctDNA; MRD; cervical carcinoma; operation; Radical radiotherapy and chemotherapy; Efficacy prediction; Recurrence monitoring
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — A total of 80 patients who meet the inclusion criteria and voluntarily sign informed consent forms are planned to be enrolled. According to the acceptable curative treatment measures of the patients, they are divided into two groups: the "operable treatment group (N=40)" and the "curative radiotherapy and chemotherapy treatment group (N=40)". Obtain tumor tissue samples from each enrolled patient (fresh tumor tissue samples (60 mg) or FFPE samples (10-15 pieces)
  Collect peripheral blood samples of 20 ml/time from multiple treatment nodes of enrolled patients, a total of 7-8 times per person
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical treatment queue (N=40): Cervical cancer patients who meet the inclusion criteria and are eligible for radical surgical resection. Collect surgical tumor tissue samples from the screening stage of patients in this queue, as well as peripheral blood samples (20 ml/time) from baseline, postoperative, postoperative radiotherapy and chemotherapy end nodes, consolidation treatment end nodes (some patients with this treatment), and multiple nodes during the 6-month follow-up stage. Perform ctDNA MRD testing in a timely manner separately
- Radical radiotherapy and chemotherapy treatment cohort (N=40): Cervical cancer patients who meet the inclusion criteria and are eligible for radical radiotherapy and chemotherapy. Collect baseline tumor tissue samples from patients during the screening phase, as well as peripheral blood samples (20 ml/time) from multiple nodes at baseline, mid-term of curative radiotherapy and chemotherapy, after curative radiotherapy and chemotherapy, after consolidation therapy (if any), and at 6 months/time during the follow-up phase. Perform ctDNA MRD testing in a timely manner separately

SUMMARY:
This study plans to enroll 80 patients with locally advanced cervical cancer (stage IB-ⅣA) confirmed by histology or cytology (according to the 2018 FIGO staging standard), who are expected to receive surgical resection or curative radiotherapy and chemotherapy. Collect baseline tumor tissue samples from patients during the treatment period, as well as peripheral blood samples (20 ml/time) from multiple treatment timepoints. Mutations in tumor tissue were detected by the 1021 genes panel, then personalized MRD monitoring probes were customized for patients, allowing for multi node peripheral blood sample ctDNA detection of enrolled patients. The clinical significance of ctDNA in prognostic stratification, recurrence monitoring, and efficacy prediction in surgical/non-surgical cervical cancer patients was explored. And compare the consistency and differences between ctDNA detection technology, imaging, and blood tumor markers in monitoring tumor disease progression, and evaluate the correlation between ctDNA status after curative treatment and patient PFS and RFS.

DETAILED DESCRIPTION:
Surgical treatment cohort (N=40):

Collect surgical tumor tissue samples from the screening stage of patients in this cohort, as well as peripheral blood samples (20 ml/time) from baseline, postoperative, postoperative radiotherapy and chemotherapy, consolidation therapy (if any), and a 2-year follow up with 6 months/time . (A total of one tissue sample, 7-8 peripheral blood samples )

Radical radiotherapy and chemotherapy treatment cohort (N=40):

Radical radiotherapy and chemotherapy cohort: Collect baseline tumor tissue samples from patients during the screening stage, as well as peripheral blood samples (20 ml/time) from baseline, mid-term of radical radiotherapy and chemotherapy, after radical radiotherapy and chemotherapy, after consolidation treatment (if any), and a 2-year follow-up stage of 6 months/time. (A total of one tissue sample, 7-8 peripheral blood samples )

If you voluntarily participate in this study, we will require your cooperation in completing the following tasks: the entire research process consists of a screening period and a follow-up period, and it will take approximately 5 years for you to complete the entire research period. If you are willing to participate in this study, we will obtain your surgical tissue samples and obtain peripheral blood samples (20 ml/time) from a total of 7-8 times during your 5-year follow-up. The MRD detection results of each timepoint throughout the entire trial process will be promptly fed back to you and your clinical doctors for your clinical treatment plan decision-making. Before formulating your clinical treatment plan, the clinical doctor will provide you with detailed information, discussion, and confirmation. Only after receiving your confirmation can you proceed with the implementation. Throughout the entire research process, we will promptly provide you with any information such as detection indicators that may affect your decision-making. You also have the right to withdraw from this study at any time without retaliation, discrimination, or any other unfair treatment. We will protect any personal privacy information of you.

If you participate in this study, you will receive a total of 6-7 free peripheral blood based deep ctDNA-MRD tests (valued at 3800 yuan/test) throughout your entire treatment and follow-up stages. Through continuous monitoring of peripheral blood ctDNA-MRD nodes, you can advance imaging to indicate your risk of disease recurrence, detect disease progression as soon as possible, effectively improve your treatment effectiveness and clinical benefits, and evaluate your treatment efficacy as soon as possible Prognosis assessment may lead to more effective control or improvement of your personal disease treatment and quality of life. The detection results of each time will be promptly fed back to you and your research doctors to assist in your clinical decision-making and disease risk warning. Meanwhile, your participation in this study may also contribute to the improvement of solid tumor diagnosis and treatment techniques, which may bring benefits to other patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* (1) Confirmed by histopathology and classified as stage IB-IVA cervical cancer patients according to the 2018 FIGO staging criteria;

  (2) Patients can receive surgical treatment or curative radiotherapy and chemotherapy;

  (3) Age range from 18 to 80 years old;

  (4) General condition: ECOG 0-2;

  (5) At least one measurable lesion (RECIST 1.1 standard);

  (6) Be able to understand the research plan and voluntarily participate in this study, and sign an informed consent form;

  (7) Good compliance, able to cooperate in collecting specimens from various nodes and provide corresponding clinical information;

  (8) Having comprehensive clinical data on imaging and pathology;

  (9) The estimated survival time of the patient is greater than 3 months;

  (10) Having sufficient organ and bone marrow functions.

Exclusion Criteria:

* 1) Within 5 years, suffering from other malignant tumors or metastatic or recurrent cervical cancer;

  (2) Has received any tumor treatment plan in the past;

  (3) Surgical resection or curative radiotherapy and chemotherapy are not acceptable;

  (4) Unable to follow the determined clinical follow-up period in conjunction with the study for follow-up;

  (5) Inability to accept or provide specified efficacy evaluation methods such as CT;

  (6) Suffering from autoimmune diseases;

  (7) Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders;

  (8) Subjects with any severe and/or uncontrolled diseases;

  (9) According to the researchers judgment, there are accompanying diseases that seriously endanger the safety of the subjects or affect the completion of the study by the subjects

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study focuses on newly diagnosed cervical cancer patients who have been confirmed by histology or cytology to undergo surgical resection or curative radiotherapy and chemotherapy in locally advanced stages (stages IB-IV). A total of 80 patients who meet the inclusion criteria and voluntarily sign informed consent forms are planned to be enrolled. According to the curative treatment measures that patients can accept, the enrolled patients are divided into a operable treatment queue (N=40) and a curative radiotherapy and chemotherapy treatment queue (N=40).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
DFS of enrolled patients for 2 years | 2 years
  DFS of enrolled patients for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Zhou, Principal Investigator — The First Affiliated Hospital of Soochow University，Director of Gynecology Department
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tian X, Ge D, Zhang F, Zhang B, Bai W, Xu X, Li Z, Cao Y, Li P, Zou K, Zou L. Dynamic analysis of circulating tumor DNA to predict prognosis and monitor therapeutic response in metastatic relapsed cervical cancer. Int J Cancer. 2021 Feb 15;148(4):921-931. doi: 10.1002/ijc.33362. Epub 2020 Nov 7. PMID 33113150
- [Background] Tian J, Geng Y, Lv D, Li P, Cordova M, Liao Y, Tian X, Zhang X, Zhang Q, Zou K, Zhang Y, Zhang X, Li Y, Zhang J, Ma Z, Shao Y, Song L, Owen GI, Li T, Liu R, Liu Q, Zou L, Zhang Z, Li Z. Using plasma cell-free DNA to monitor the chemoradiotherapy course of cervical cancer. Int J Cancer. 2019 Nov 1;145(9):2547-2557. doi: 10.1002/ijc.32295. Epub 2019 Apr 16. PMID 30919951
- [Background] Pan Y, Zhang JT, Gao X, Chen ZY, Yan B, Tan PX, Yang XR, Gao W, Gong Y, Tian Z, Liu SM, Lin H, Sun H, Huang J, Liu SY, Yan HH, Dong S, Xu CR, Chen HJ, Wang Z, Li P, Guan Y, Wang BC, Yang JJ, Tu HY, Yang XN, Zhong WZ, Xia X, Yi X, Zhou Q, Wu YL. Dynamic circulating tumor DNA during chemoradiotherapy predicts clinical outcomes for locally advanced non-small cell lung cancer patients. Cancer Cell. 2023 Oct 9;41(10):1763-1773.e4. doi: 10.1016/j.ccell.2023.09.007. PMID 37816331
- [Background] Zhang JT, Liu SY, Gao W, Liu SM, Yan HH, Ji L, Chen Y, Gong Y, Lu HL, Lin JT, Yin K, Jiang BY, Nie Q, Liao RQ, Dong S, Guan Y, Dai P, Zhang XC, Yang JJ, Tu HY, Xia X, Yi X, Zhou Q, Zhong WZ, Yang XN, Wu YL. Longitudinal Undetectable Molecular Residual Disease Defines Potentially Cured Population in Localized Non-Small Cell Lung Cancer. Cancer Discov. 2022 Jul 6;12(7):1690-1701. doi: 10.1158/2159-8290.CD-21-1486. PMID 35543554
- [Background] Liu T, Yao Q, Jin H. Plasma Circulating Tumor DNA Sequencing Predicts Minimal Residual Disease in Resectable Esophageal Squamous Cell Carcinoma. Front Oncol. 2021 May 20;11:616209. doi: 10.3389/fonc.2021.616209. eCollection 2021. PMID 34094900
- [Background] Schwarzenbach H, Hoon DS, Pantel K. Cell-free nucleic acids as biomarkers in cancer patients. Nat Rev Cancer. 2011 Jun;11(6):426-37. doi: 10.1038/nrc3066. Epub 2011 May 12. PMID 21562580
- [Background] Azad TD, Chaudhuri AA, Fang P, Qiao Y, Esfahani MS, Chabon JJ, Hamilton EG, Yang YD, Lovejoy A, Newman AM, Kurtz DM, Jin M, Schroers-Martin J, Stehr H, Liu CL, Hui AB, Patel V, Maru D, Lin SH, Alizadeh AA, Diehn M. Circulating Tumor DNA Analysis for Detection of Minimal Residual Disease After Chemoradiotherapy for Localized Esophageal Cancer. Gastroenterology. 2020 Feb;158(3):494-505.e6. doi: 10.1053/j.gastro.2019.10.039. Epub 2019 Nov 9. PMID 31711920
- [Background] Xu JZ, Wen F, Wang XR. The eIF3a Arg803Lys genetic polymorphism is associated with susceptibility to and chemoradiotherapy efficacy in cervical carcinoma. Kaohsiung J Med Sci. 2017 Apr;33(4):187-194. doi: 10.1016/j.kjms.2017.01.008. Epub 2017 Mar 13. PMID 28359406
- [Background] Beharee N, Shi Z, Wu D, Wang J. Diagnosis and treatment of cervical cancer in pregnant women. Cancer Med. 2019 Sep;8(12):5425-5430. doi: 10.1002/cam4.2435. Epub 2019 Aug 6. PMID 31385452
- [Background] Lagheden C, Eklund C, Lamin H, Kleppe SN, Lei J, Elfstrom KM, Sundstrom K, Andrae B, Sparen P, Dillner J. Nationwide comprehensive human papillomavirus (HPV) genotyping of invasive cervical cancer. Br J Cancer. 2018 May;118(10):1377-1381. doi: 10.1038/s41416-018-0053-6. Epub 2018 Mar 21. PMID 29559733
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338